CLINICAL TRIAL: NCT06395142
Title: Changes of Plantar Pressure and Electroencephalographic Signals During Pedal Walking and Vision-deprivation Walking in Stroke Patients.
Brief Title: Plantar Pressure and Electroencephalographic Signals During Pedal and Vision-deprived Walking in Stroke Patients.
Status: Completed | Type: Observational
Sponsor: Geriatric Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jing Zhao, Principal Investigator, Geriatric Hospital of Nanjing Medical University
Other Study IDs: LL2024018-1
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: Electroencephalography; pedal walking; visual deprivation; challenging task
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke participants: Stroke participants performe pedal walking and visual-deprivation walking successively.
  Interventions: Other: pedal walking; Other: visual-deprivation walking

INTERVENTIONS:
Other: pedal walking — Pedal walking is a challenging task for stroke participants and can be used as a means of stroke rehabilitation. A cross-sectional study is conducted to investigate the real-time changes in plantar pressure and electroencephalogram during pedal walking in stroke participants.
Other: visual-deprivation walking — visual-deprivation walking is a challenging task for stroke participants and can be used as a means of stroke rehabilitation.A cross-sectional study is conducted to investigate the real-time changes in plantar pressure and electroencephalogram during visual-deprivation walking in stroke participants.

SUMMARY:
Complex task training may be more effective than simple task training in promoting functional recovery and brain restructuring in stroke participants. The researchers intend to investigate the real-time changes in plantar pressure and electroencephalographic signals in stroke participants during two complex tasks: pedal walking and visual-deprivation walking. The research hypothesis is that pedal walking and visual-deprivation walking can improve the difference of plantar pressure between the affected and unaffected lower limbs of stroke participants, and cause corresponding electroencephalographic changes.

DETAILED DESCRIPTION:
Stroke participants perform the following tasks after wearing a plantar pressure device and a 32-lead electroencephalographic cap. First, stroke participants walk on the pedal on the lower limbs of the affected side. Then the researchers cover the participants' eyes with an eye mask, the participants perform the task of visual-deprivation walking. Finally, the participants walk on a flat surface. Each walking task lasts for 60 seconds. The participants can rest for 3-5 minutes between tasks.

ELIGIBILITY:
Inclusion Criteria:

* MRI or CT diagnosis of the first stroke onset；
* The onset of the stroke occurred more than 30 days;
* Safely walk 50 meters without assistance.

Exclusion Criteria:

* Cerebellar injury；
* Brain stem injury；
* Visual impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke participants recruited from inpatient and outpatient departments of tertiary hospitals.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
phase-amplitude coupling | Real-time monitoring of electroencephalography data will occur while participants are walking. The Time Frame for data collection will encompass the entire duration of each participant's walking session, which lasts for 60 seconds.
  Phase-amplitude coupling is a type of cross-phase coupling that represents the coupling between the phase of slow oscillations and the amplitude of fast oscillations.
phase-frequency coupling | Real-time monitoring of electroencephalography data will occur while participants are walking. The Time Frame for data collection will encompass the entire duration of each participant's walking session, which lasts for 60 seconds.
  Phase-frequency coupling is a generic form of the cross-frequency coupling model, representing the coupling between the slow oscillations phase and the fast oscillations frequency.
phase-phase coupling | Real-time monitoring of electroencephalography data will occur while participants are walking. The Time Frame for data collection will encompass the entire duration of each participant's walking session, which lasts for 60 seconds.
  Phase-phase coupling is a special form of cross-phase coupling that represents the coupling between the phases of slow and fast oscillations, which can occur even when the coupling is very weak.
Amplitude-amplitude coupling | Real-time monitoring of electroencephalography data will occur while participants are walking. The Time Frame for data collection will encompass the entire duration of each participant's walking session, which lasts for 60 seconds.
  Amplitude-amplitude coupling is a form of cross-phase coupling that represents the coupling between the amplitudes of slow oscillations and fast oscillations .
relative power | Real-time monitoring of electroencephalography data will occur while participants are walking. The Time Frame for data collection will encompass the entire duration of each participant's walking session, which lasts for 60 seconds.
  Relative power reflects the frequency domain changes of electroencephalogram.
weight Phase Lag Index | Real-time monitoring of electroencephalography data will occur while participants are walking. The Time Frame for data collection will encompass the entire duration of each participant's walking session, which lasts for 60 seconds.
  The weight phase lag index is an index of brain functional connectivity, can continuously measure the connectivity of the coupling of neural oscillatory activity.
peak pressure | Through study completion, an average of 2 months.
  Peak pressure reflects the maximum pressure on the entire sole of the foot.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Li Zhang, doctor, Study Chair — Geriatric Hospital of Nanjing Medical University
Locations (1):
- Geriatric Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliveira AS, Schlink BR, Hairston WD, Konig P, Ferris DP. Restricted vision increases sensorimotor cortex involvement in human walking. J Neurophysiol. 2017 Oct 1;118(4):1943-1951. doi: 10.1152/jn.00926.2016. Epub 2017 Jul 5. PMID 28679843
- [Background] Fettrow T, Hupfeld K, Tays G, Clark DJ, Reuter-Lorenz PA, Seidler RD. Brain activity during walking in older adults: Implications for compensatory versus dysfunctional accounts. Neurobiol Aging. 2021 Sep;105:349-364. doi: 10.1016/j.neurobiolaging.2021.05.015. Epub 2021 May 31. PMID 34182403
- [Result] Krakauer JW. Motor learning: its relevance to stroke recovery and neurorehabilitation. Curr Opin Neurol. 2006 Feb;19(1):84-90. doi: 10.1097/01.wco.0000200544.29915.cc. PMID 16415682